CLINICAL TRIAL: NCT06698523
Title: Evaluation of Bubble-Blower Exercise and Pin-Wheel Exercise on Dental Anxiety in Children: A Randomized Controlled Trial
Brief Title: To Assess Breathing Exercise as a Relaxation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Passant Mohamed Ibrahim Attia Elbahy, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PED23-4M
Record Dates: First submitted 2024-11-05; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Dental Anxiety
Keywords: breathing exercise; play toys; heart rate; venham picture test; salivary alpha amylase
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tell- show-Do (No Intervention): Control group
- Bubble-blower (Experimental): breathing exercise technique using bubble-blower
  Interventions: Behavioral: Breathing exercise
- Pin-wheel (Experimental): breathing exercise technique using Pin-wheel
  Interventions: Behavioral: Deep breathing

INTERVENTIONS:
Behavioral: Breathing exercise — bubble blower used as play toys to facilitate the breathing exercise
  Other Names: bubble blower exercise
  Arms: Bubble-blower
Behavioral: Deep breathing — pin wheel used as a play toy for achievement of breathing exercise
  Arms: Pin-wheel

SUMMARY:
in this study investigator evaluate the effectiveness of breathing exercise using two different play toys in reducing dental anxiety.

DETAILED DESCRIPTION:
bubble blower and pin wheel are used to facilitate breathing exercise and to reduce dental anxiety hence more cooperation of participants during dental treatment

ELIGIBILITY:
Inclusion Criteria:

* children that had been introduced to dental setting without receiving any dental treatment
* According to Corah 's dental anxiety scale children classified with score 19 or more
* No learning disability or psychological disorder or parental anxiety

Exclusion Criteria:

* children in emergency visit
* Allergy to anesthetic drugs
* Use of analgesic before treatment
* Teeth with necrotic pulp
* children whose parents refused to sign informed consent

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Heart rate to assess child's dental anxiety | during dental treatment after local anesthetic injection. Heart rate is measured in beats/min measured twice, first before any dental treatment and measured a second time after 7-10 minutes after injection of local anesthesia
  correlating participants anxiety to heart rate the higher the heart rate indicating the higher the anxiety level of patients
Venham picture test used to assess dental anxiety | during dental treatment recorded before any treatment is done and after five minutes of injection of local anesthesia
  score 0-8, it is an eight cards photos that are shown to children if child chooses the more anxious child in picture this is recorded as a score, the higher the score the more anxious the participants.
Salivary Alpha amylase | before any dental treatment is done and 7-10 minutes after injection of local anesthesia
  collecting saliva sample for assessment of alpha amylase by ELISA test, saliva collected twice before and after injection of local anesthesia and correlating concentration to dental anxiety the higher the concentration of alpha amylase indicates more anxious children

SECONDARY OUTCOMES:
Innovation of a new protocol in behavior management prior to painful dental procedure | during dental treatment that will take 15-30 minutes
  breathing exercise using play toys as behavior management

CONTACTS AND LOCATIONS:
Overall Officials: Passant Elbahy, Principal Investigator — Ain Shams University Faculty of Dentistry
Locations (1):
- Ain Shams University Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No